CLINICAL TRIAL: NCT03047681
Title: Tryptase Levels as a Marker of Mast Cell Activity and the Prognostic Implication in Patients Post Transcatheter Aortic Valve Replacement
Brief Title: Tryptase Level as a Marker of Complications in Transcatheter Aortic Valve Replacement
Acronym: TAVR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0678-15-TLV
Record Dates: First submitted 2017-02-08; First posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Transcatheter Aortic Valve Implantation Prosnosis and Complications
Keywords: TAVR; tryptse; mast

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tryptase level in serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: patients undergoin transcatheter aortic valve implantation
  Interventions: Diagnostic Test: venous blood withdrawl
- Control group: patient undergoing diagnostic coronary angiography
  Interventions: Diagnostic Test: venous blood withdrawl

INTERVENTIONS:
Diagnostic Test: venous blood withdrawl — patients will be asked for a venous blood sample

SUMMARY:
An association between mast cells and outcomes of patients undergoing transcatheter aortic valve replacement (TAVR) has not been studied to our knowledge. We aim to characterize tryptase levels dynamics during TAVR; Demonstrate whether tryptase level post-TAVR can be used as a prognostic marker.

DETAILED DESCRIPTION:
Inflammation is known to have a detrimental effect on outcome of patients with myocardial infarction (MI) [1, 2] as well as reperfusion injury (RI) [3]. Previous trials have shown correlation between the extent of an inflammatory response and postoperative complications and worse outcomes in patients undergoing cardiac surgery [4, 5, 6, 7] including valve replacement [8]. Transcatheter aortic valve replacement (TAVR) may be associated with inflammation [5, 9] as well. A few possible mechanisms may be responsible, such as tissue injury due to mechanical trauma, vascular complications, and possible suboptimal organ perfusion due to bleeding, ventricular pacing, balloon valvuloplasty, deployment, post-dilatation, or repositioning of the valve prosthesis [10]. Accumulating data show that peri-procedural inflammation is associated with worse outcomes and complications of TAVR [11, 12, 13, 14, 15], and may predict increased mortality in patients after TAVR [16, 17, 18, 19, 20].

Inflammation is a complex process and includes many types of cells including mast cells. The association between mast cells, as part of the inflammatory process, and RI has been thoroughly studied. Mast cells have been linked to RI in many organs [21], contributing to insult to the myocardium. This association has been suggested from animal models [22, 23, 24] as well as recent human trials which showed that tryptase, an abundant protease found in mast cell granules, is elevated in ST segment elevation myocardial infarction (STEMI) patients treated with primary percutaneous coronary intervention (PCI) [25].

Therefore, it is reasonable to assume that mast cells may have a role in the inflammation process involved in patients undergoing TAVR. Moreover, such association with mast cells may be used to predict adverse outcomes.

To our knowledge, an association between mast cells and outcomes of patients undergoing TAVR has not been studied.

METHODS Peripheral venous blood from 30 patients undergoing TAVR will be withdrawn to examine tryptase levels, as a marker of mast cell activity. Blood samples will be taken at 0 hours (before the procedure) and a second sample will be taken up to 2 hours post-procedure.

CRP will be examined in each patient pre and post TAVR. Tryptase levels will be examined in 10 patients undergoing diagnostic coronary angiography.

PRIMARY OBJECTIVE We aim to: 1. Characterize tryptase levels dynamics during TAVR 2. Demonstrate whether tryptase level post-TAVR can be used as a prognostic marker.

Primary outcome - mortality at 1 year Secondary outcomes - Major complications at 7 days and 30 days, including death, major stroke, acute kidney injury, paravalvular regurgitation, permanent pacemaker implantation, coronary artery obstruction, heart block, vascular injury, pericardial hemorrhage.

REFERENCES:

1. Patel MR, Mahaffey KW, Armstrong PW, Weaver WD, Tasissa G, Hochman JS, Todaro TG, Malloy KJ, Rollins S, Theroux P, Ruzyllo W, Nicolau JC, Granger CB. Prognostic usefulness of white blood cell count and temperature in acute myocardial infarction (from the CARDINAL Trial). Am J Cardiol 2005;95:614-618.
2. Theroux P, Armstrong PW, Mahaffey KW, Hochman JS, Malloy KJ, Rollins S, Nicolau JC, Lavoie J, Luong TM, Burchenal J, Granger CB. Prognostic significance of blood markers of inflammation in patients with ST-segment elevation myocardial infarction undergoing primary angioplasty and effects of pexelizumab, a C5 inhibitor: a substudy of the COMMA trial. Eur Heart J 2005;26:1964-1970.
3. Ibáñez B, Heusch G, Ovize M, Van de Werf F. Evolving therapies for myocardial ischemia/reperfusion injury. J Am Coll Cardiol. 2015 Apr 14;65(14):1454-71.
4. Cremer J, Martin M, Redl H, Bahrami S, Abraham C, Graeter T, Haverich A, Schlag G, Borst HG. Systemic inflammatory response syndrome after cardiac operations. Ann Thorac Surg 1996;61:1714-1720.
5. Lindman BR, Goldstein JS, Nassif ME, Zajarias A, Novak E, Tibrewala A, Vatterott AM, Lawler C, Damiano RJ, Moon MR, Lawton JS, Lasala JM, Maniar HS. Systemic inflammatory response syndrome after transcatheter or surgical aortic valve replacement. Heart 2015 Apr;101(7):537-45.
6. Kilger E, Heyn J, Beiras-Fernandez A, et al. Stress doses of hydrocortisone reduce systemic inflammatory response in patients undergoing cardiac surgery without cardiopulmonary bypass. Minerva Anestesiol. 2011;77:268-274.
7. Clarizia NA, Manlhiot C, Schwartz SM, et al. Improved outcomes associated with intraoperative steroid use in high-risk pediatric cardiac surgery. Ann Thorac Surg. 2011;91(4):1222-1227.
8. Prat C, Ricart P, Ruyra X, et al. Serum concentrations of procalcitonin after cardiac surgery. J Card Surg. 2008;23(6):627-632.
9. Stähli BE1, Grünenfelder J, Jacobs S, Falk V, Landmesser U, Wischnewsky MB, Lüscher TF, Corti R, Maier W, Altwegg LA. Assessment of inflammatory response to transfemoral transcatheter aortic valve implantation compared to transapical and surgical procedures: a pilot study. J Invasive Cardiol. 2012 Aug;24(8):407-11.
10. Sinning JM1, Scheer AC, Adenauer V, Ghanem A, Hammerstingl C, Schueler R, Müller C, Vasa-Nicotera M, Grube E, Nickenig G, Werner N. Systemic inflammatory response syndrome predicts increased mortality in patients after transcatheter aortic valve implantation. Eur Heart J. 2012 Jun;33(12):1459-68.
11. Masson JB1, Kovac J, Schuler G, Ye J, Cheung A, Kapadia S, Tuzcu ME, Kodali S, Leon MB, Webb JG. Transcatheter aortic valve implantation: review of the nature, management, and avoidance of procedural complications. JACC Cardiovasc Interv. 2009 Sep;2(9):811-20.
12. Toggweiler S1, Webb JG. Challenges in transcatheter aortic valve implantation. Swiss Med Wkly. 2012 Dec 17;142:w13735.
13. Rettig TC1, Rigter S1, Nijenhuis VJ2, van Kuijk JP2, ten Berg JM2, Heijmen RH3, van de Garde EM4, Noordzij PG. The systemic inflammatory response syndrome predicts short-term outcome after transapical transcatheter aortic valve implantation. J Cardiothorac Vasc Anesth. 2015 Apr;29(2):283-7.
14. Krumsdorf U1, Chorianopoulos E, Pleger ST, Kallenbach K, Karck M, Katus HA, Bekeredjian R. C-reactive protein kinetics and its prognostic value after transfemoral aortic valve implantation. J Invasive Cardiol. 2012 Jun;24(6):282-6.
15. Van Linden A1, Kempfert J, Rastan AJ, Holzhey D, Blumenstein J, Schuler G, Mohr FW, Walther T. Risk of acute kidney injury after minimally invasive transapical aortic valve implantation in 270 patients. Eur J Cardiothorac Surg. 2011 Jun;39(6):835-42; discussion 842-3.
16. Zahn R, Gerckens U, Grube E, Linke A, Sievert H, Eggebrecht H, Hambrecht R, Sack S, Hauptmann KE, Richardt G, Figulla HR, Senges J. Transcatheter aortic valve implantation: first results from a multi-centre real-world registry. Eur Heart J 2011;32:198-204
17. Sinning JM, Ghanem A, Steinhauser H, Adenauer V, Hammerstingl C, Nickenig G, Werner N. Renal function as predictor of mortality in patients after percutaneous transcatheter aortic valve implantation. JACC Cardiovasc Interv 2010;3:1141-1149.
18. Nuis RJ, van Mieghem NM, Tzikas A, Piazza N, Otten AA, Cheng J, van Domburg RT, Betjes M, Serruys PW, de Jaegere PP. Frequency, determinants and prognostic effects of acute kidney injury and red blood cell transfusion in patients undergoing transcatheter aortic valve implantation. Catheter Cardiovasc Interv 2011;77:881-889.
19. Aregger F, Wenaweser P, Hellige GJ, Kadner A, Carrel T, Windecker S, Frey FJ. Risk of acute kidney injury in patients with severe aortic valve stenosis undergoing transcatheter valve replacement. Nephrol Dial Transplant 2009;24:2175-2179.
20. Bagur R, Webb JG, Nietlispach F, Dumont E, De Larochelliere R, Doyle D, Masson JB, Gutierrez MJ, Clavel MA, Bertrand OF, Pibarot P, Rodes-Cabau J. Acute kidney injury following transcatheter aortic valve implantation: predictive factors, prognostic value, and comparison with surgical aortic valve replacement. Eur Heart J 2010;31:865-874. Van Linden A, Kempfert J, Rastan AJ, Holzhey D, Blumenstein J, Schuler G, Mohr FW, Walther T. Risk of acute kidney injury after minimally invasive trans-apical aortic valve implantation in 270 patients. Eur J Cardiothorac Surg 2011;39:835-42.
21. Yang MQ1, Ma YY, Ding J, Li JY. The role of mast cells in ischemia and reperfusion injury. Inflamm Res. 2014 Nov;63(11):899-905.
22. Masini E, Giannella E, Bianchi S, Mannaioni PF: Histamine and lactate dehydrogenase (LDH) release in ischemic myocardium of the guinea-pig. Agents Actions 1987;20:281-283.
23. Masini E1, Bianchi S, Gambassi F, Palmerani B, Pistelli A, Carlomagno L, Mannaioni PF. Ischemia reperfusion injury and histamine release in isolated and perfused guinea-pig heart: pharmacological interventions. Agents Actions. 1990 Apr;30(1-2):198-201
24. Frangogiannis NG1, Perrard JL, Mendoza LH, Burns AR, Lindsey ML, Ballantyne CM, Michael LH, Smith CW, Entman ML. Stem cell factor induction is associated with mast cell accumulation after canine myocardial ischemia and reperfusion. Circulation. 1998 Aug 18;98(7):687-98.
25. Shaomin Chen, Di Mu, Ming Cui, Chuan Ren, Shu Zhang, Lijun Guo, and Wei Gao. Dynamic changes and clinical significance of serum tryptase levels in STEMI patients treated with primary PCI. Biomarkers. 2014 Nov;19(7):620-4.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Capable of giving informed consent
* Undergoing TAVR

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients who undergo TAVR
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-02 (Estimated); Primary Completion 2017-08-01 (Estimated); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 1 year
  mortality

SECONDARY OUTCOMES:
Mortality | 7 and 30 days
  mortality at 7 and 30 days
Complications | 30 days
  Post procedural complications - major stroke, acute kidney injury, paravalvular regurgitation, permanent pacemaker implantation, coronary artery obstruction, heart block, vascular injury, pericardial hemorrhage

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
Only the principle investigator will have access to IPD